CLINICAL TRIAL: NCT06757803
Title: The Analgesic Effect of Retro-laminar Block Versus Paravertebral Block in Patients With Multiple Fracture Ribs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Aboelyosr, Demonstrator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLB VS PVB fracture ribs
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Rib Fracture
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): patients will be subjected to rertrolaminar block
  Interventions: Procedure: rertrolaminar block
- group 2 (Experimental): patients will be subjected to paravertebral block
  Interventions: Procedure: paravertebral block

INTERVENTIONS:
Procedure: rertrolaminar block — Positioning
  The patient is positioned in a lateral decubitus position with the affected side up. The patient's arm on the affected side is placed behind the head. The patient's spine is aligned and the shoulder is elevated to expose the paravertebral space.
  *Ultrasound imaging
  A high-frequency linear ultrasound probe (5-12 MHz) is placed in a paramedian sagittal plane at the desired level of block. The probe is oriented so that the transverse processes are visualized on the lateral side of the screen and the vertebral laminae are visualized on the medial side of the screen. The interlaminar space is visualized as a hypoechoic region between the laminae.
  *Needle insertion
  A short bevel block needle (20-22 G) is inserted through the skin at the caudal end of the ultrasound probe, aiming cephalad. The needle is advanced under real-time ultrasound guidance until the tip of the needle contacts the lamina. The needle is then slightly withdrawn and the local anesthetic is injected into t
  Arms: group 1
Procedure: paravertebral block — * Patient Preparation
  * Place the patient in the lateral decubitus position with the side of the block facing up.
  * Position the patient's arm so that it is resting comfortably on the operating table.
  * Prepare the skin over the block site with an antiseptic solution.
  * Sterilely drape the area.
  * Ultrasound Imaging
  * Place the ultrasound probe in a transverse plane at the level of the desired block.
  * Identify the following anatomical landmarks:
  * Vertebral body
  * Transverse process
  * Pleura
  * Intercostal space
  * Needle Insertion
  Use a sterile ultrasound-guided needle. Insert the needle in-plane from a lateral to medial direction, aiming for the apex of the paravertebral space.
  The needle should be advanced until it is just beyond the transverse process.
  *Test Aspiration
  Aspirate to ensure that the needle is not in a blood vessel.
  * Local Anesthetic Injection
  * Inject the local anesthetic slowly, aspirating frequently.
  * The local anesthetic should be injected int
  Arms: group 2

SUMMARY:
Rib fractures are a common injury, occurring in up to 10% of all trauma patients. Multiple rib fractures can be particularly painful and debilitating, making it difficult for patients to breathe and cough. This can lead to complications such as atelectasis, pneumonia, and respiratory failure.

Adequate pain control is essential for patients with rib fractures. This can help to improve respiratory function, reduce the risk of complications, and speed up recovery.

Paravertebral block (PVB) is a regional anaesthetic technique that is commonly used for pain management in patients with rib fractures. It involves injecting local anaesthetics into the paravertebral space, which is a region of tissue located between the transverse processes of the vertebrae and the pleura. PVB is an effective way to block the sensory nerves that supply the thoracic region, including the ribs.

However, PVB can be technically challenging to perform, and there is a risk of complications such as pneumothorax and pleural puncture.

Retrolaminar block (RLB) is a newer regional anaesthetic technique that has been proposed as an alternative to PVB for pain management in patients with rib fractures. RLB involves injecting local anaesthetics into the retrolaminar space, which is a region of tissue located between the lamina of the vertebra and the epidural space.

RLB is thought to be easier to perform than PVB, and there is a lower risk of complications. However, there is limited studies support the use of RLB for pain management in patients with rib fractures.

The primary objective of this research is to compare the analgesic efficacy of retrolaminar block (RLB) and paravertebral block (PVB) in patients with fracture ribs.

Secondary objectives include:

* To compare the safety of RLB and PVB
* To compare the duration of analgesia provided by RLB and PVB

DETAILED DESCRIPTION:
Rib fractures are a common injury, occurring in up to 10% of all trauma patients. Multiple rib fractures can be particularly painful and debilitating, making it difficult for patients to breathe and cough. This can lead to complications such as atelectasis, pneumonia, and respiratory failure.

Adequate pain control is essential for patients with rib fractures. This can help to improve respiratory function, reduce the risk of complications, and speed up recovery.

Paravertebral block (PVB) is a regional anaesthetic technique that is commonly used for pain management in patients with rib fractures. It involves injecting local anaesthetics into the paravertebral space, which is a region of tissue located between the transverse processes of the vertebrae and the pleura. PVB is an effective way to block the sensory nerves that supply the thoracic region, including the ribs.

However, PVB can be technically challenging to perform, and there is a risk of complications such as pneumothorax and pleural puncture.

Retrolaminar block (RLB) is a newer regional anaesthetic technique that has been proposed as an alternative to PVB for pain management in patients with rib fractures. RLB involves injecting local anaesthetics into the retrolaminar space, which is a region of tissue located between the lamina of the vertebra and the epidural space.

RLB is thought to be easier to perform than PVB, and there is a lower risk of complications. However, there is limited studies support the use of RLB for pain management in patients with rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* * Age 18 years or older

  * American Society of Anesthesiologists (ASA) physical status I-III
  * Rib fractures, as confirmed by X-ray or computed tomography (CT) scan
  * Both sexes, males and females.

Exclusion Criteria:

* *Patient refusal.

  * Infection at the injection site
  * Allergy to local anesthetics
  * Neurological deficit
  * Spinal deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
total post operative analgesic consumption | 48 hours
  total analgesic consumption in 1st 48hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kotze A, Scally A, Howell S. Efficacy and safety of different techniques of paravertebral block for analgesia after thoracotomy: a systematic review and metaregression. Br J Anaesth. 2009 Nov;103(5):626-36. doi: 10.1093/bja/aep272. PMID 19837806